CLINICAL TRIAL: NCT02003742
Title: Efficacy and Safety of a Single Transrectal Ultrasound(TRUS)-Guided Intraprostatic Injection of NX-1207 in Patients With Lower Urinary Tract Symptoms Associated With Benign Prostatic Hyperplasia: A Phase III European Study
Brief Title: Efficacy and Safety of a Single TRUS-guided Intraprostatic Injection of NX-1207 in Patients With LUTS Due to BPH
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped because in two other clinical studies the drug was not superior in comparison with placebo
Sponsor: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NX1207-IT-CL 0414
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2022-05-26 (Actual); Status verified 2013-12

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: LUTS; BPH
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — fexapotide; Tamsulosin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- NX-1207 (Experimental): Subjects randomised to the NX-1207 group will receive a single NX-1207 (2.5 mg) TRUS-guided intraprostatic injection (under antibiotic prophylaxis), followed by a placebo QD oral treatment for 12 months.
  Interventions: Drug: NX-1207
- Comparator (Active Comparator): Subjects randomised to the comparative arm will undergo TRUS only (under placebo prophylaxis) and will continue the tamsulosin 0.4 mg QD oral treatment for 12 months
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: NX-1207 — Single TRUS-guided intraprostatic injection of 2.5 mg of NX-1207
  Arms: NX-1207
Drug: Tamsulosin — 1 film coated, prolonged release tablet of tamsulosin 0.4 mg, to be taken orally (p.o.) QD
  Arms: Comparator

SUMMARY:
The purpose of the this international, multicenter, randomised, single-blind, parallel group, Phase III study is to demonstrate that a single transrectal ultrasound (TRUS)-guided intraprostatic injection of NX-1207 provides a long lasting therapeutic improvement of Lower Urinary Tract Symptoms (LUTS) associated with Benign Prostatic Hyperplasia (BPH) in patients not adequately controlled by medical therapy with α-blockers, as assessed by a change from baseline in the International Prostate Symptom Score (IPSS) total score.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Age 45 or older;
* Medical history of LUTS/BPH
* Use of a marketed α-blocker for LUTS/BPH in the last 8 weeks;
* LUTS/BPH not adequately controlled by medical therapy with α-blockers;
* Presence of moderate-severe LUTS (IPSS ≥ 15) at screening and at baseline (after a 4 week run-in period with tamsulosin 0.4 mg QD);
* Prostate Volume ≥ 30 mL and ≤ 70 mL (as assessed by TRUS);
* Qmax < 15 mL/sec based on a minimum void of 125 mL;
* Agree not to use any other approved or experimental BPH or overactive bladder (OAB) medication anytime during the core study;
* Agree to perform follow-up visits even in case of oral treatment discontinuation before study end;
* Satisfactory compliance to run-in medication at Visit 2 (baseline).

Exclusion Criteria:

* Previous surgical or invasive prostate treatments such as TURP, TUMT, TUNA, laser or any other minimally invasive treatment;
* Acute or chronic prostatitis or suspected prostatitis including chronic pain, intermittent pain or abnormal sensation in the penis, testis, anal or pelvic area in the past 12 months;
* PSA ≥ 10 ng/mL. In case of a PSA between 4.0 and 10.0 ng/mL, prostate cancer must have been ruled out to the satisfaction of the clinical Investigator by an historical biopsy;
* Prostate or bladder cancer, history of pelvic irradiation;
* Active or recurrent urinary tract infections (more than 1 episode in the last 12 months);
* History of neurogenic bladder or LUTS secondary to neurologic disease;
* Use of self-catheterization for urinary retention;
* Post-void residual urine volume > 200 mL;
* Haematuria which has not been appropriately evaluated to determine safe subject participation;
* Renal insufficiency (serum creatinine >2.0 mg/dL);
* Liver insufficiency (any liver function tests [LFTs]>2x upper limit of normal [ULN]);
* Poorly controlled diabetes (type 1 or type 2), as determined by HbA1c >6% and/or glycosuria;
* Any bleeding disorder such as haemophilia, clotting factor(s) deficiency or bleeding diathesis;
* Immunosuppressive disorders, such as Human Immunodeficiency (HIV) Virus, Acquired Immune Deficiency Syndrome (AIDS), lymphoproliferative disorders;
* Acute or chronic intestinal disease, such as ulcerative colitis, Crohn's disease, acute gastroenteritis in the run-in period; acute painful perianal disorder;
* Unstable cardiovascular or cerebrovascular disease (including acute myocardial infarction, unstable angina pectoris, by-pass, Percutaneous Transluminal Coronary Angioplasty (PTCA), congestive heart failure NYHA Class III-IV, stroke, transient ischemic attack and episodes of cardiac arrhythmia requiring treatment in the last 6 months);
* Any condition that would interfere with the subject's ability to provide informed consent, to comply with study instructions, or that might confound the interpretation of the study results, such as dementia, psychosis, manic depressive disorder, post-traumatic stress disorder, stroke, Alzheimer's, depression, psychiatric illness, history or current evidence of drug or alcohol abuse within the last 12 months etc.;
* Participation in a study of any investigational drug or device within the previous 6 months;
* Hypersensitivity or contraindication to tamsulosin use;
* Use of prohibited medications that could endanger subjects performing the intraprostatic injection or that could interfere with the evaluation of study parameters;
* Men planning to have children in the future;
* Any other condition that may interfere with the study or endanger the subject.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-09; Primary Completion 2015-01-29 (Actual); Study Completion 2015-01-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the total IPSS score. | 12 months
  The primary efficacy parameter is the change from baseline in the total score (Questions 1 to 7) of the IPSS at 12 months.
  The IPSS questionnaire will be filled by the subjects in blind conditions and will be reviewed by the investigators for its completeness. Validated local translations of the IPSS questionnaire will be used in each country.

SECONDARY OUTCOMES:
Effects on Lower Urinary Tract Symptoms | 1,3,6,9 and 12 months
  * Change from baseline in IPSS total score at 1, 3, 6 and 9 months;
  * Change from baseline in IPSS subscores for storage symptoms;
  * Change from baseline in IPSS subscores for voiding symptoms;
  * Response rate by IPSS
Effects on Quality of Life (QoL) due to urinary symptoms | 1,3,6,9 and 12 months
  * Change from baseline in IPSS subscore Quality of Life due to urinary symptoms;
  * Change from baseline in BPH Impact Index
Effects on general health related Quality of Life | 12 months
  The change from baseline in the EQ-5D-5L questionnaire at 12 months or in case of early termination will be considered.
  The EQ-5D-5L questionnaire is a standardised validated instrument for use as a measure of health outcome.
Patient's global assessment of treatment | 12 months
  A patient-rated global assessment of treatment benefit, satisfaction and willingness to continue will be performed at 12 months (or in case of early termination) by using the BSW questionnaire.
  The BSW is a validated questionnaire that consists of three, single-item measures designed to capture the patient's perception of the effect of treatment in terms of the relative benefit, their satisfaction, and their intention or willingness to continue on therapy.
Effects on maximum urinary flow rate (Qmax) | 3,6,9 and 12 months
  To evaluate the effect on urinary flow, the change from baseline in maximum urinary flow (Qmax) at 3, 6, 9, 12 months will be considered. The same validated device and procedure will be used in all centres and a blinded centralized reading is foreseen.
Effects on prostate volume | 3 and 12 months
  The change from baseline in TRUS assessed prostate volume at 3 and 12 months (or in case of early termination) will be considered.

OTHER OUTCOMES:
Long term follow-up evaluation | 24 months
  The following data will be evaluated:
  * Percentage of subjects requiring medical therapy, MIST, TURP or surgery for LUTS/BPH and time to treatment failure;
  * Change from baseline in the total score of the IPSS;
  * Change from baseline in QoL due to urinary symptoms
  * Change from baseline in general health-related QoL (EQ-5D-5L);
  * SAEs and episodes of acute urinary retention.

CONTACTS AND LOCATIONS:
Locations (5):
- Klinikum der Ludwig-Maximilians-universität München, Munich, Germany
- Vita e Salute University, Department of Urology, Istituto Scientifico Ospedale San Raffaele, Milan, Italy
- Niepubliczny Zaklad Opieki Zdrowotnej Specjalista, Kutno, Poland
- Hospital General Universitario Gregorio Marañón, Madrid, Spain
- Sheffield Teaching Hospitals NHS Foundation Trust, Royal Hallamshire Hospital, Sheffield, United Kingdom